CLINICAL TRIAL: NCT06986850
Title: FeelSync: Tailoring Ecological Momentary Assessments and Interventions for Emotion Awareness, Regulation, and Mental Health Outcomes
Acronym: FeelSync
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marta Marciniak (Other)
Responsible Party: Sponsor-Investigator, Marta Marciniak, Assistant Professor, Erasmus University Rotterdam
Organization: Erasmus University Rotterdam (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: ETH2425-0653
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Stress
Keywords: ecological momentary assessment; ecological momentary intervention; language; cognitive reappraisal; emotion regulation; emotion awareness; mental health
MeSH Terms: conditions — Language; Emotional Regulation; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Ecological Momentary Assessment with self-generated emotion description (Active Comparator): Ecological Momentary Assessment with participant's self-generated emotion description in an open-ended question form, in English, provided five times daily for seven consecutive days
  Interventions: Device: Ecological Momentary Assessment mobile application
- Ecological Momentary Assessment with pre-defined set of emotion items to select (Active Comparator): Ecological Momentary Assessment with pre-defined set of emotion items to select in a multiple-choice question form, in English, provided five times daily for seven consecutive days
  Interventions: Device: Ecological Momentary Assessment mobile application
- Ecological Momentary Assessment with pre-defined set of emotion items to rate on a Likert scale (Active Comparator): Ecological Momentary Assessment with pre-defined set of emotion items to rate on a seven-point Likert scale, in a slider form, in English, provided five times daily for seven consecutive days
  Interventions: Device: Ecological Momentary Assessment mobile application
- Ecological Momentary Intervention with self-generated emotion description (Experimental): Ecological Momentary Intervention focused on cognitive reappraisal, with a possibility to choose between distancing and positive reappraisal, provided three times daily and preceded by Ecological Momentary Assessment with participant's self-generated emotion description in an open-ended question form, in English, provided five times daily for seven consecutive days
  Interventions: Device: FeelSync mobile application
- Ecological Momentary Intervention with self-generated emotion description in mother tongue (Experimental): Ecological Momentary Intervention focused on cognitive reappraisal, with a possibility to choose between distancing and positive reappraisal, provided three times daily and preceded by Ecological Momentary Assessment with participant's self-generated emotion description in an open-ended question form, in participant's mother tongue, provided five times daily for seven consecutive days
  Interventions: Device: FeelSync mobile application
- Ecological Momentary Intervention with pre-defined set of emotion items to select (Experimental): Ecological Momentary Intervention focused on cognitive reappraisal, with a possibility to choose between distancing and positive reappraisal, provided three times daily and preceded by Ecological Momentary Assessment with pre-defined set of emotion items to rate on a seven-point Likert scale, in a slider form, in English, provided five times daily for seven consecutive days
  Interventions: Device: FeelSync mobile application
- Ecological Momentary Intervention with pre-defined set of emotion items to rate on a Likert scale (Experimental): Ecological Momentary Intervention focused on cognitive reappraisal, with a possibility to choose between distancing and positive reappraisal, provided three times daily and preceded by Ecological Momentary Assessment with pre-defined set of emotion items to rate on a seven-point Likert scale, in a slider form, in English, provided five times daily for seven consecutive days
  Interventions: Device: FeelSync mobile application

INTERVENTIONS:
Device: FeelSync mobile application — Ecological Momentary Intervention focused on cognitive reappraisal for distressing autobiographical memories, with a possibility to choose between distancing and positive reappraisal.
  Arms: Ecological Momentary Intervention with pre-defined set of emotion items to rate on a Likert scale; Ecological Momentary Intervention with pre-defined set of emotion items to select; Ecological Momentary Intervention with self-generated emotion description; Ecological Momentary Intervention with self-generated emotion description in mother tongue
Device: Ecological Momentary Assessment mobile application — Ecological Momentary Assessment used for self-monitoring of emotional states.
  Arms: Ecological Momentary Assessment with pre-defined set of emotion items to rate on a Likert scale; Ecological Momentary Assessment with pre-defined set of emotion items to select; Ecological Momentary Assessment with self-generated emotion description

SUMMARY:
This study investigates how different ways of reflecting on emotions in daily life influence emotional awareness, emotion regulation, and mental health. Using the FeelSync mobile app over the course of seven days, participants are prompted multiple times a day to report on their current emotional state in various formats (e.g., rating scales, multiple choice, or free text). In some groups, participants also receive brief daily exercises designed to help them practice cognitive reappraisal-a strategy that involves reframing stressful situations to reduce their emotional impact. The study aims to assess not only the overall effectiveness of these reappraisal exercises but also whether the type of emotional self-report used before the intervention affects its impact. All participants complete questionnaires before and after the app phase to track changes in mood, stress, emotional awareness, and regulation.

ELIGIBILITY:
Inclusion Criteria:

* Owning a smartphone
* Proficiency in English language
* Being a student
* Age between 18 to 30 years old

Exclusion Criteria:

- Severe mental health disorder

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 490 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Baseline (pre-intervention, study day 1) and Follow-up (post intervention, study day 9)
  Self-report questionnaire, Range: 0 - 40 Higher scores: Worse outcome (higher perceived stress)
Beck Depression Inventory II | Baseline (pre-intervention, study day 1) and Follow-up (post intervention, study day 9)
  Self-report questionnaire, Range: 0 - 63 Higher scores: Worse outcome (more severe depressive symptoms)
State-Trait Anxiety Inventory | Baseline (pre-intervention, study day 1) and Follow-up (post intervention, study day 9)
  Self-report questionnaire, [state scale only], Range: 20 - 80 Higher scores: Worse outcome (greater state anxiety)
Emotion Regulation Questionnaire | Baseline (pre-intervention, study day 1) and Follow-up (post intervention, study day 9)
  Self-report questionnaire, Reappraisal subscale: Range 1 - 7 (mean of 6 items) Higher scores: Better outcome (more frequent use of cognitive reappraisal) Suppression subscale: Range 1 - 7 (mean of 4 items) Higher scores: Worse outcome (more frequent use of suppression)
Cognitive Emotion Regulation Questionnaire | Baseline (pre-intervention, study day 1) and Follow-up (post intervention, study day 9)
  Self-report questionnaire, Subscale range: 2 - 10 per strategy
  Higher scores:
  On adaptive strategies (e.g., positive reappraisal, putting into perspective): Better outcome On maladaptive strategies (e.g., rumination, catastrophizing): Worse outcome
Toronto Alexithymia Scale | Baseline (pre-intervention, study day 1) and Follow-up (post intervention, study day 9)
  Self-report questionnaire, Range: 20 - 100 Higher scores: Worse outcome (greater difficulties in identifying and describing feelings; lower emotional awareness)

SECONDARY OUTCOMES:
Mobile Agnew Relationship Measure | Follow-up (post intervention, study day 9)
  Self-report questionnaire, Range: 16-112 Higher scores: Better outcome (stronger perceived therapeutic alliance with the app/intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Rotterdam, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Only anonymized data from the self-report questionnaires will be shared via Open Science Framework.
Supporting Information: Analytic Code
Time Frame: 09/2025-09/2035
Access Criteria: Anyone will be able to access anonymized participant data from self-report questionnaires.